CLINICAL TRIAL: NCT05529485
Title: Research and Quantification of Factors Influencing Endothelial Damage During Phacoemulsification
Brief Title: Quantification of Factors Influencing Endothelial Damage During Phacoemulsification
Acronym: PREDICSPILOT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-11Obs-CHRMT
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Endothelial Cell Loss, Corneal; Cataract; Phacoemulsification
MeSH Terms: conditions — Corneal Endothelial Cell Loss; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cataract surgery by phacoemulsification — Cataract surgery by phacoemulsification

SUMMARY:
The aim of this study is to determine the principal factors that influence endothelial cell loss three month post cataract surgery.

Methods: Multi center observational Cohort study, inclusion period from 12/01/2022 to 10/06/2022. One hundred and seventy-five eyes of hundred and four patients who have appointment for cataract surgical indication were included. The percentage of corneal endothelial cell loss was quantified using specular microscopy before and 3 months after the surgery.

14 variables (pre-operative and intra-operative) that could be associated to endothelial cell injury were selected.

A bivariate analysis of relationship between these factors and endothelial cell loss at 3 months was performed by simple linear regression (Wilcoxon and Fischer tests). Multivariate analysis was performed by multiple linear regression in order to identify the factors independently related to endothelial cell loss.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cataract surgery
* Visual acuity monoyer scale <8/10e (> +0.2 logMar)
* Nuclear, cortical and posterior subcapsular cataract with normal density to severe in the LOCSIII classification
* Covered by the social security scheme
* Have given their oral agreement

Exclusion Criteria:

* Corneal disease: keratitis, dystrophy or corneal degeneration
* Any disease of the anterior segment
* Low preoperative endothelial cell density <1000 c/mm²
* Pregnancy, lactation
* Risk factors for surgical per-operative complication
* Uncontrolled ocular pressure
* Combined surgery (cataract with corneal graft, cataract with glaucoma surgery, cataract with vitrectomy, ....)
* Under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
The difference in central corneal endothelial cell density (cells/mm²) between the 1st preoperative measurement and the postoperative measurement at 3 months. | 3 months after cataract surgery
  Specular counts were performed by the orthoptists, residents or physicians of the department using a Nidek CEM-530 specular microscope with automated central cell counting without corneal contact. Three measurements were performed at each consultation and the average of these three measurements was reported.

SECONDARY OUTCOMES:
Postoperative visual acuity | 3 months after cataract surgery
  best spectacle corrected visual acuity is evaluated using Monoyer scale, scores ranging from 1 to 10, higher scores mean a better outcome; score 10 is the best.
Postoperative corneal edema | 3 months after cataract surgery
  Corneal edema is measured using specular microscope with pachymeter

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc Perone, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (1):
- CHR Metz-Thionville/Hopital de Mercy, Metz, France